CLINICAL TRIAL: NCT04466475
Title: A Phase I Trial Evaluating Escalating Doses of 211At-Labeled Anti-CD38 Monoclonal Antibody (211At-OKT10-B10) Combined With Melphalan as Conditioning Prior to Autologous Hematopoietic Cell Transplantation for Patients With Multiple Myeloma
Brief Title: Radioimmunotherapy (211At-OKT10-B10) and Chemotherapy (Melphalan) Before Stem Cell Transplantation for the Treatment of Multiple Myeloma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: NIH terminated funding. Study was closed before any participants were enrolled.
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1006317; NCI-2019-06979 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10306 (Other: Fred Hutch/University of Washington Cancer Consortium); R01CA205248 (NIH)
Record Dates: First submitted 2020-07-08; First posted 2020-07-10 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-09

CONDITIONS: Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (211At-OKT10-B10, melphalan, PBSC transplantation) (Experimental): Patients receive 211At-OKT10-B10 IV continuously on day -10 to day - 4 (approximately day -7) and melphalan via infusion on day -2. Patients then undergo HCT on day 0.
  Interventions: Biological: Astatine At 211 Anti-CD38 Monoclonal Antibody OKT10-B10; Drug: Melphalan; Procedure: Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: Astatine At 211 Anti-CD38 Monoclonal Antibody OKT10-B10 — Given IV
  Other Names: 211At-OKT10-B10; [211At]OKT10-B10; Astatine 211-labeled Anti-CD38 Monoclonal Antibody OKT10-B10; Astatine At 211 Anti-CD38 MoAb OKT10-B10; Astatine-211-OKT10-B10; At211-OKT10-B10
Drug: Melphalan — Given via infusion
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo PBSC transplantation
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation

SUMMARY:
This phase I trial studies the side effects and best dose of 211At-OKT10-B10 when given together with melphalan before a stem cell transplantation in treating patients with multiple myeloma. The radioimmunotherapy drug 211At-OKT10-B10 is a monoclonal antibody, called OKT10-B10, linked to a radioactive substance called 211At. OKT10-B10 attaches to CD38 positive cancer cells in a targeted way and delivers 211At to kill them. Drugs used in chemotherapy, such as melphalan, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving 211At-OKT10-B10 with melphalan before a stem cell transplant may kill more cancer cells.

DETAILED DESCRIPTION:
OUTLINE: This is a dose-escalation study of 211At-OKT10-B10.

Patients receive 211At-OKT10-B10 intravenously (IV) continuously on day -10 to day - 4 (approximately day -7) and melphalan via infusion on day -2. Patients then undergo hematopoietic cell transplantation (HCT) on day 0.

After completion of study treatment, patients are followed for 30 days, between 80 and 90 days, at 6, 9, 12, 18, and 24 months, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of multiple myeloma
* Patients must have autologous hematopoietic stem cells collected with a minimum CD34+ stem cell yield of >= 4 x 10^6 CD34+ cells/kg of body weight
* Subjects must have disease meeting criteria for clinical relapse or progressive disease (International Myeloma Working Group [IMWG] consensus criteria) and a history of >= 1 prior autologous stem cell transplant(s)
* Subjects must have received at least 3 prior lines of therapy: an immunomodulatory drug, a proteasome inhibitor, and a CD38-targeting antibody

  * Aline of therapy is defined as one or more cycles of a planned treatment program. This may consist of one or more planned cycles of a single-agent therapy or combination therapy, as well as a sequence of treatments administered in a planned manner. For example, a planned treatment approach of induction therapy followed by autologous stem cell transplantation, followed by maintenance is considered one line of therapy. A new line of therapy starts when a planned course of therapy is modified to include other treatment agents (alone or in combination) as a results of disease progression, relapse, or toxicity. A new line of therapy also starts when a planned period of observation off therapy is interrupted by a need for additional treatment for the disease
* Subjects must have an estimated creatinine clearance greater than 60 ml per minute by the following formula (Cockcroft-Gault). Serum creatinine value must be within 28 +/- days prior to registration
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) score =< 2 or Karnofsky score >= 70%
* Ability to provide informed consent
* Subjects 18 years of age

Exclusion Criteria:

* Subjects with a history of plasma cell leukemia
* History of central nervous system involvement by multiple myeloma
* Prior radioimmunotherapy or radiation of > 20 Gy to pelvis or at maximally tolerated levels to any critical normal organ
* Prior allogeneic hematopoietic cell transplant
* More than 2 prior autologous hematopoietic cell transplants
* Subjects with medullary or extramedullary plasmacytoma/s measuring > 3 cm by magnetic resonance imaging (MRI) or positron emission tomography (PET)-computed tomography (CT) (radiated lesions are exempt from this criterion)
* Subjects with a history of any one of the following cardiovascular conditions within the past 6 months: Class III or IV heart failure as defined by the New York Heart Association (NYHA), cardiac angioplasty or stenting, myocardial infarction, unstable angina, or other clinically significant cardiac disease as determined by the principal investigator (PI) or designee
* Subjects with corrected QT (QTc) prolongation at baseline
* Subjects with a history of cardiac arrhythmia and a heart rate > 100 beats per minute (BPM) (oral beta-blocker [excluding sotalol] and/or calcium channel blocker therapy are acceptable to achieve rate control)
* History of reactive airway disease and clinically significant asthma requiring any form of medical treatment in the prior three months
* Left ventricular ejection fraction < 40%
* Corrected diffusing capacity of the lungs for carbon monoxide (DLCO) < 50% or receiving supplemental continuous oxygen
* Liver abnormalities: fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction as evidenced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis, or symptomatic biliary disease.
* Bilirubin > 2 times the upper limit of normal
* Aspartate aminotransferase [AST] and alanine aminotransferase [ALT] > 2 times the upper limit of normal
* Subjects who are known to be seropositive for human immunodeficiency virus (HIV)
* Women of childbearing potential who are pregnant (beta-human chorionic gonadotropin [HCG]+) or breast feeding
* Fertile subjects unwilling to use contraceptives during and for 12 months post-transplant
* Subjects with untreated and uncontrolled infection at time of enrollment
* Subjects with known amyloid light-chain (AL) subtype amyloidosis
* Known allergy to murine-based monoclonal antibodies
* Known contraindications to radiotherapy
* History of another primary malignancy that has not been in remission for at least 2 years (the following are exempt from the 2-year limit: non-melanoma skin cancer, curatively treated localized prostate cancer, and cervical carcinoma in situ on biopsy or a squamous intraepithelial lesion on Papanicolaou [PAP] smear)
* Any anti-CD38 monoclonal antibody within 30 days of anticipated date of infusion of 211At-OKT10-B10
* Individuals with a history of CTCAE grade 4 gastrointestinal toxicity associated with prior high-dose melphalan conditioning therapy (previous autologous stem cell transplant)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-27 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | Up to 30 days post-transplant
  Defined a true dose limiting toxicity (DLT) probability of 25% of subjects, where a DLT is defined as any grade 3-5 nonhematologic regimen-related toxicity within the first 30 days following autologous hematopoietic cell transplantation.

SECONDARY OUTCOMES:
Achievement of response | Between days +80 to +90 post-transplant
  Measured per the International Myeloma Working Group criteria. The response rates (partial response [PR] or better) will be estimated along with the exact 95% confidence interval.
Duration of response | From response (PR or better) to disease relapse or death, assessed up to 5 years
  Duration of response will be estimated using Kaplan-Meier methodology.
Overall survival | From transplantation to death, assessed up to 2 years post-transplant
  Kaplan-Meier methodology will be used to estimate the 2-year overall survival.
Progression-free survival | From transplantation to disease relapse or death, assessed up to 2 years post-transplant
  Kaplan-Meier methodology will be used to estimate the 2-year progression-free survival.
Rates of minimal residual disease (MRD) | At days 28, and +80 to +90 post-transplant
  MRD will be assessed using multi-color flow cytometry and next generation sequencing in conjunction with functional imaging (i.e., positron emission tomography-computed tomography). The proportion who achieve MRD will be estimated along with an exact 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Damian J. Green, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No